CLINICAL TRIAL: NCT06975345
Title: Short, Medium and Long Term Effects of a Protocol of Hip Flexor Stretching, Exercise and Pain Managment Education, Function and Disability in Patients With Chronic, Mechanical, Non-specific Low Back Pain. Randomized Controlled Clinical Trial.
Brief Title: Effects of a Protocol of Hip Flexor Stretching on Chronic Mechanical, Non-specific LBP.
Acronym: HipFlexinCLBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Universidad de Zaragoza (Other); Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Aleksander Kucza, MSc, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AWFWroclawUNIZAR.PhDAlek
Record Dates: First submitted 2025-04-25; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Pain; Musculoskeletal Manipulations; Low Back Pain, Mechanical
Keywords: manual therapy,; spine,; low back pain,; Chronic Low Back Pain,; Muscle Stretching Exercises,; Range of Motion, Articular,; Body composition,; Numeric Pain Rating Scale (NPRS)
MeSH Terms: conditions — Pain; Low Back Pain | interventions — Educational Status; Dosage Forms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Participants will receive a protocol of hip flexors stretching, exercise and education for chronic low back pain added to the standard of care in the Polish public health services prescribed by the medicine doctor.
  Interventions: Other: Multicomponent intervention. Hip flexors stretching, Strengthening exercises and education and medical treatment (Medication and medical counselling); Drug: Medical treatment.
- Control group (Active Comparator): Participants will receive only the standard of care in the Polish public health services prescribed by a medicine doctor.
  Interventions: Drug: Medical treatment.

INTERVENTIONS:
Other: Multicomponent intervention. Hip flexors stretching, Strengthening exercises and education and medical treatment (Medication and medical counselling) — Hip flexors stretching (Adaptation from Evjenth and Hamberg)
  Strengthening Exercise
  * Deep squats
  * Flexo-extension of the ankle on a step over the head of metatarsal bones
  * Plank
  * Strengthening knee flexors and hip extensors
  * Lunges with a stick behind the patient back
  Education Pain relieving positions identified will be taught to the patient to use when they feel their pain.
  Identifying and learning to avoid pain positions or activities that increase pain.
  When the pain occur self stretching of hip flexors on the couch or the chair must be done
  Arms: Experimental group
Drug: Medical treatment. — A medical doctor will prescribe the treatment following the standard of care in Polish public health services. Treatment will consist of medication and counseling.

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of a stretching, exercise and education protocol versus usual care in improving pain, function and disability in patients with non-specific mechanical chronic low back pain (CLBP). The research hypothesis is: A combination of hip flexors stretching, exercise and education is more effective than usual care to improve pain, function and disability in patients with CLBP.

Participants will be randomly allocated in one of the two treatment groups. Pain, function and disability will be assessed before starting treatment, after the end of the treatment and one month , three months and one year after the end of the treatment.

DETAILED DESCRIPTION:
Study design: the study is a randomized controlled study that will be conducted in a physiotherapy center in Poland. Potential subjects will be identified in public and private health services by a medicine doctor who will be responsible for screening subjects for eligibility and enrolling into the study.

Men and Women between 18 and 75 years old that will fulfill the criteria and will sign the informed consent will be randomly assigned to one of the two treatment groups. Randomization will be 1:1 ratio and the method to generate random allocation will be a random computer generated numbers table.

Evaluator, outcome assessor, will be blinded to the participant's group assignment.

The study has been approved by the research ethics committee of Wroclaw University of Health Sciences and Sports. The study will be conducted in accordance with ethical principles of the declaration of Helsinki (75th World Medical Association General Assembly , Helsinki, Finland, October 2024)

Treatment Groups:

Experimental group: Participants will receive a protocol of hip flexors stretching, exercise and education for chronic low back pain added to the standard of care in the Polish public health services prescribed by the medicine doctor.

Control group: Participants will receive only the standard of care in the Polish public health services prescribed by a medicine doctor.

The treatment period will consist of two weeks. Experimental group will receive 3 treatment sessions during this period of time. Control group will receive medication and counsels under medical doctor criteria.

The patients will be assessed at baseline (t0), after the treatment period (t1), 1 month after the end of the treatment (t2), three months after the end of the treatment (t3), and one year after the end of the treatment (t4).The variables that will be collected will be: Pain (NPRS), function (ROM), disability (ODI) and other descriptive and sociodemographic variables.

Statistical analysis will be performed to describe the sample, groups and comparison between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Medical diagnosis of chronic, mechanical, non-specific pain in the lumbar spine (M54, M51) - chronic low back pain.
* Obtaining written consent to conduct research
* Must be able to swallow tablets

Exclusion Criteria:

* Pregnancy
* Pacemaker
* Active cancer
* To consent to conduct research
* Difficulty communicating
* The presence of a metal plate in the head and metal screws in the body
* Condition after operations in the area of the lumbar spine
* Condition after fractures in the lumbar spine
* Contraindications to manual therapy or exercise
* Has participated in a lumbar spine exercise or manual therapy program in the last three months
* Present clear signs of having suffered a significant lumbar injury
* Inability to maintain standing or a supine or prone position
* No possibility to perform the stretching of hip flexors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline, to complete the treatments, on average 2 weeks, 1, 3 and 12 months after the end of treatment
  Numeric Pain Rating Scale (NPRS) The NPRS will be used to ask the patient about the level of pain that he/she feels considering from 0 to 10, where 0 represents the absence of pain and 10 represents the most intense pain, used to measure the pain experienced by the patient. The participant will answer the NPRS, responding to the average, maximum and minimum pain experienced throughout its duration.

SECONDARY OUTCOMES:
Lumbar Range of Motion | Baseline, to complete the treatments, on average 2 weeks, 1 month after the end of treatment.
  The MyoMotion( Noraxon, USA) is a device used to measure degrees of range of motion (ROM) in the lumbar spine. It consists of accelerometers and a program. The range of flexion, extension, will be measured in degrees.
ROM in Thomas test | Baseline,to complete the treatments, on average 2 weeks, 1 month after the end of treatment
  The MyoMotion( Noraxon, USA) is a device used to measure degrees of range of motion (ROM) in the lumbar spine. It consists of accelerometers and a program. The range of flexion, extension, will be measured in degrees.
Clinical Measure of extension. | Baseline, to complete the treatments, on average 2 weeks, 1 month after the end of treatment.
  To assess a patient's ability to extend their spine, a clinical method will be used and recorded. This method involves asking the patient how far they can reach while looking at a measuring tape.
Anatomical distribution of pain | Baseline, to complete the treatments, on average 2 weeks, 1, 3 and 12 months after the end of treatment
  Patients will draw on a body silhouette the region where they feel pain.
ROM in Straight Leg Raise Test | Baseline, to complete the treatments, on average 2 weeks, 1 month after the end of treatment.
  Range of motion (ROM) in a straight leg raise (SLR) test that measures the hip's flexibility while putting tension on the sciatic nerve. The test helps diagnose nerve root compression in the lower lumbar spine. Measures range of motion of the hip.
Quality of Life level | Baseline, to complete the treatments, on average 2 weeks, 1, 3 and 12 months after the end of treatment
  The SF-36 questionnaire includes 8 multi-item subscales assessing social functioning, mental health, vitality, physical functioning, role limitations due to physical problems, role limitations due to emotional problems, pain, and general health perception. The total score ranges from 0 to 100, with a higher score indicating a better health-related quality of life.
Kinesiophobia | Baseline, to complete the treatments, on average 2 weeks, 1, 3 and 12 months after the end of treatment
  The Tampa Scale of Kinesiophobia (TSK) is a 17-item self-report questionnaire that measures fear of movement or re-injury. It's used to identify people with chronic pain who have high levels of fear of movement.
Degree of Functional Disability | Baseline,to complete the treatments, on average 2 weeks, 1, 3 and 12 months after the end of treatment
  Oswestry Disability Index ( ODI) a questionnaire that measures how much disability someone has in their daily lives. It's used to assess low back pain. It assesses 10 activities of daily living, including pain, walking, sleeping, and social life. The ODI score ranges from 0-100, with 0 being the best and 100 being the worst.
Physical activity level | Baseline, to complete the treatments, on average 2 weeks, 1, 3 and 12 months after the end of treatment
  Measured using the short version of the International Physical Activity Questionnaire (IPAQ). Questionnaire contains 7 questions about all types of physical activity related to everyday life, work and leisure. Results are reported in categories depending on the variable 'MET minutes a week'. MET minutes represent the amount of energy expended carrying out physical activity. High physical activity (one hour or more of physical activity per day), moderate physical activity (half an hour of physical activity per day) or low physical activity (not meeting any of the criteria for either moderate or high levels of physical activity).
Body composition analysis | Baseline
  Body mass (Body composition analyzer BC 418 MA by Tanita), body height (height gauge SECA 217), based on them, determination of the BMI index and BMI percentile using percentile grids developed based on the OLAF program. Analysis of general and segmental parameters:
  FatP - body fat mass in %, FatM - body fat mass in kg, FFM - body fat-free mass, TBW - body water quantity in kg and %. FFF index - based on the values of body fat and fat-free tissue, the general and segmental fat-free index is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehasport Wroclaw, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided